CLINICAL TRIAL: NCT00307229
Title: A Phase I Trial Investigating the Safety and Immunogenicity of an Adenovirus Encoding Rat HER-2 Administered Intradermally to Patients With Metastatic or Locally Recurrent Breast Cancer
Brief Title: Adenovirus Encoding Rat HER-2 in Patients With Metastatic Breast Cancer (AdHER2.1)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Ontario Clinical Oncology Group (OCOG) (Other)
Collaborators: Ontario Cancer Research Network (Network); Canadian Breast Cancer Research Alliance (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CTA-Control-100643
Record Dates: First submitted 2006-03-24; First posted 2006-03-27 (Estimated); Last update posted 2012-06-04 (Estimated); Status verified 2012-05

CONDITIONS: Metastatic Breast Cancer; Recurrent Breast Cancer
Keywords: metastatic breast cancer; recurrent breast cancer
MeSH Terms: conditions — Breast Neoplasms

INTERVENTIONS:
Biological: adenoviral vector encoding rat Her-2/neu — Group 1 1 x 10'7 pfu (2.5 X 10'6 pfu per injection site)(1.6 x 10'9 particles) Group 2 5 x 10'7 pfu (1.25 X 10'7 pfu per injection site)(8.0 x10'9 particles) Group 3 1 x 10'8 pfu (5 x 10'7 pfu per injection site)(1.6 x10'10 particles)

SUMMARY:
To determine the maximum tolerated dose and/or maximum attainable dose of a vaccine consisting of adenovector expressing rat Her-2/neu in patients with metastatic or locally recurrent breast cancer.

ELIGIBILITY:
Inclusion Criteria:

1. metastatic or locally recurrent breast cancer,
2. 18 years of age or older,
3. Her-2/neu positive (3+ by immunohistochemistry or FISH +),
4. One of the following

   1. currently receiving hormonal therapy or are candidates for such or,
   2. being considered for trastuzumab or,
   3. their cancer has progressed on trastuzumab

Exclusion Criteria:

1. Pregnant or lactating women.
2. Prior or concurrent malignancies except treated basal cell or squamous carcinoma of the skin or in situ cancer of the cervix or any other cancer treated and presumed cured more than five years prior to study entry.
3. Currently receiving chemotherapy, immunotherapy, adenoviral gene therapy or biological cancer therapy. [Note: concurrent hormonal therapy (tamoxifen,aromatase inhibitors, or megace) is permitted.].
4. Treatment with trastuzumab within 4 weeks prior to first dose of vaccine therapy.
5. Hemoglobin < 80 g/L or granulocytes < 1.5 x 109 /L or lymphocytes < 1.0 x 109 /L or platelets < 100 x 109 /L.
6. Baseline liver enzymes (AST or ALT) greater than 3 times upper limit of normal or greater than 5 times upper limit of normal if liver metastases present and/or bilirubin greater than 50 mmol.
7. CD4 cells < 0.5 x 109 /L
8. Patients with documented brain metastases.
9. Patients with any acute illness that would interfere with vaccination
10. Any patients requiring concurrent immunosuppressive therapy (e.g. corticosteroids).
11. Eastern Cooperative Oncology Group (ECOG) performance status of > 2.
12. Patients with a life expectancy of less than 6 months.
13. Geographic inaccessibility which would preclude follow-up. Patients registered on the trial must be treated and followed at the Jewish General Hospital.
14. Failure to give written informed consent.
15. Baseline left ventricular ejection fraction (LVEF) < 55% by echocardiography or MUGA scan.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2006-03; Primary Completion 2009-07 (Actual); Study Completion 2012-05 (Actual)

PRIMARY OUTCOMES:
toxicity | Weeks 4, 6, 7, 10, 14, 18, 22, 26

SECONDARY OUTCOMES:
tumour response | Weeks 6, 18

CONTACTS AND LOCATIONS:
Overall Officials: Gerry Batist, M.D., Study Chair — Lady Davis Institute for Medical Research Jewish General Hospital; Ronan Foley, M.D., Principal Investigator — Hamilton Health Sciences Corporation; Mark Levine, M.D., Principal Investigator — Ontario Clinical Oncology Group (OCOG)
Locations (1):
- Sir Mortimer B. Davis - Jewish General Hospital, Montreal, Quebec, Canada